CLINICAL TRIAL: NCT01949805
Title: A Randomized, Open-label, Multicenter, Controlled, Parallel Arm, Phase III Study Assessing the Efficacy and Safety of AOP2014 vs. Hydroxyurea in Patients With Polycythemia Vera
Brief Title: Pegylated Interferon Alpha-2b Versus Hydroxyurea in Polycythemia Vera
Acronym: PROUD-PV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Collaborators: PharmaEssentia (Co-Sponsor for USA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROUD-PV; 2012-005259-18 (EudraCT Number)
Record Dates: First submitted 2013-09-06; First posted 2013-09-25 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — peginterferon alfa-2b; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyurea (Active Comparator): Hydroxyurea capsules (500 mg each). Daily intake of doses from 500 mg Q2D to 3000 mg QD
  Interventions: Drug: Hydroxyurea
- Peg-P-IFN-alpha-2b (AOP2014) (Experimental): Peg-P-IFN-alpha-2b at 50mcg to max 500 mcg, given every other week as one subcutanous injection
  Interventions: Drug: Peg-P-IFN-alpha-2b (AOP2014)

INTERVENTIONS:
Drug: Peg-P-IFN-alpha-2b (AOP2014) — Pegylated interferon alpha 2b given Q2W as SC injection
  Other Names: AOP2014; P1101
  Arms: Peg-P-IFN-alpha-2b (AOP2014)
Drug: Hydroxyurea — Hydroyurea capsules taken daily po
  Other Names: HU; Hydroxycarbamide; brand name Litalir (or other)
  Arms: Hydroxyurea

SUMMARY:
Phase III study to compare the efficacy and safety of the novel monopegylated interferon alpha 2b AOP2014 versus Hydroxyurea (the current licensed therapy for this disease). One year treatment of patients with polycythemia vera. Objective is to demonstrate non-inferiority of AOP2014 vs. HU in terms of disease response rate in both HU naïve and currently treated patients, diagnosed with Polycythemia Vera. Response is measured as normalisation of key lab parameters as well as normalized spleen size.

DETAILED DESCRIPTION:
Hydroxyurea is an established first-line treatment option currently approved in several European countries for Polycythemia Vera (PV) patients requiring a cytoreductive therapy (Barbui et al, 2011). Clinical trials have shown that HU is an effective drug for preventing thrombosis in PV compared to phlebotomy (Michiels et al, 1999).

The main concern of a long term treatment with HU is its potential leukaemogenicity: based on the mechanism of action, HU can potentially accelerate the accumulation of mutations in DNA and increase the risk of leukaemic transformation (Dingli et Tefferi, 2006). However, there is currently no clear clinical data to confirm leukaemogenicity of HU in patients with PV (Tefferi, 2012).

Even though IFN-alpha has shown its activity in PV in the 1980s, it is still considered as an experimental treatment in Europe due to pending approval in this indication (Barbui et al, 2011). It induces major or complete molecular remissions in patients with PV accompanied by a reduction in the risk of thrombosis and bleeding - the major determinants of morbidity in this indication (Hasselbalch, 2011). However, only low doses are tolerated and significant adverse effects from long-term use may limit its usefulness.

Pegylated interferons are better tolerated and are the preferred options of treatment in PV patients (Kiladjian et al, 2008) despite the lack of evidences based on well-designed randomized controlled clinical studies.

AOP2014 is a next generation pegylated interferon (Peg-P-IFN-alpha-2b), with the addition of proline in the N-terminal end.

AOP2014 like all interferon suppresses the malignant clone causing PV and subsequently is expected to possibly defer the onset of or avoid long term sequelae of PV. In addition, a reduction in the frequency of phlebotomies should be achieved. The peg-P-IFN-alpha-2b might potentially have a positive impact on reducing the drop-out rate compared to conventional IFNs. It is expected that the reduced frequency of administration of AOP2014 will contribute to higher compliance rates.

The maximum tolerated dose as well as the safety, efficacy and pharmacokinetics of AOP2014 were assessed in a phase I/II study in patients with PV. After 24 evaluable patients had entered the Phase I dose finding part, the MTD was defined at the level of 540 µg administered every two weeks. Another 27 patients were recruited in order to further investigate the drug efficacy and safety in PV. Efficacy results of AOP2014 were promising. By visit 18, 53.0% of the patients had reached complete response (12 evaluable patients). Adverse events were manageable and rarely necessitated treatment discontinuation.

AOP2014 was shown to have a prolonged plasma half-life with a concomitant increase in AUC. This is expected to enhance the therapeutic window of peg-IFN-alpha-2b.

The safety profile of type I interferons alpha is believed to be well characterized after clinical experience for nearly 20 years. Since the dose is carefully titrated to the optimal effective dose no additional risks for the patients are expected. HU, the IMP-comparator in the study, is the standard reference treatment in PV.

This phase III study was designed to compare, for the first time, the efficacy and safety of HU with a pegylated prolin-interferon alpha-2b (AOP2014) in patients with PV. Two populations will be assessed: HU naïve patients and patients currently treated or pre-treated with HU for less than 3 years, not responding to HU treatment (according to criteria in this protocol).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Diagnosis of Polycythemia Vera according to the WHO 2008 criteria (Barbui et al, 2011) with the mandatory presence of JAK2V617F mutation as the major disease criterion.
3. For previously cytoreduction untreated patients - documented need of cytoreductive treatment

   - leukocytosis (WBC>10G/L for two measurements within one week)
4. For patients currently treated or pre-treated with HU, all of the following criteria:

   * being non responders (as defined by the response criteria for primary endpoint)
   * total HU treatment duration shorter than three years
   * no documented resistance or intolerance as defined by modified Barosi et al, 2009 criteria
5. Hospital Anxiety and Depression Scale (HADS) score 0-7 on both subscales
6. Patients with HADS score of 8-10 inclusive on either or both of the subscales may be eligible following psychiatric assessment that excludes clinical significance of the observed symptoms in the context of potential treatment with an interferon alpha
7. Signed written informed consent

Exclusion Criteria:

1. Any systematic cytoreduction for PV prior study entry with exception of HU for shorter than 3 years (see respective inclusion criterion)
2. Any contraindication to any of the IMPs (pegylated interferon or hydroxyurea) or their excipients
3. Any systemic exposure to a non-pegylated or pegylated interferon alpha
4. Documented autoimmune disease at screening or in the medical history
5. Clinically relevant pulmonary infiltrates, pneumonia, and pneumonitis at screening
6. Systemic infections, e.g. hepatitis B, hepatitis C, or HIV at screening
7. Known PV-related thromboembolic complications in the abdominal area (e.g. portal vein thrombosis, Budd-chiari syndrome) and/or splenectomy in the medical history
8. Any investigational drug less than 6 weeks prior to the first dose of study drug or not recovered from effects of prior administration of any investigational agent
9. History or presence of depression requiring treatment with antidepressant
10. HADS score equal to or above 11 on either or both of the subscales
11. Any risk of suicide at screening or previous suicide attempts
12. Any significant morbidity or abnormality which may interfere with the study participation
13. Pregnancy and breast-feeding females of reproductive potential and males not using effective means of contraception
14. History of active substance or alcohol abuse within the last year
15. Evidence of severe retinopathy (e.g. cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension)
16. Thyroid dysfunction not adequately controlled
17. Patients tested positively with TgAb and / or TPOAb at screening
18. History of major organ transplantation
19. History of uncontrolled severe seizure disorder
20. Leukocytopenia at the time of screening
21. Thrombocytopenia at the time of screening
22. History of malignant disease, including solid tumours and hematological malignancies (except basal cell and squamous cell carcinomas of the skin and carcinoma in situ of the cervix that have been completely excised and are considered cured) within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Disease response rate | Month 12
  Disease response rate is defined as hematocrit <45% without phlebotomy (at least 3 months since last phlebotomy), platelets <400 G/L, leukocytes <10 G/L , and normal spleen size

SECONDARY OUTCOMES:
Disease response | at month 3, 6 and 9
JAK2 allelic burden changes | at month 6 and 12
time to response | from inclusion until first response confirmation
  will be measured during the study period of 12 months
duration of response | during the 12 months of study duration
  from the first documented response on study
number of phlebotomies | from inclusion until month 12
blood parameters | from inclusion until month 12
  biweekly
spleen size | at month 3, 6, 9 and 12
  both centrally (blinded assessment) and locally
disease related symptoms | from inclusion until month 12
  biweekly
adverse events | from inclusion until month 12
  biweekly
protocol-specific adverse events of special interest | from inclusion until month 12
  biweekly

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Gisslinger, MD, Principal Investigator — Medical University of Vienna
Locations (58):
- Austria (7):
  - LKH Graz, Graz
  - University Hospital Innsbruck, Innsbruck
  - Elisabethinen Hospital Linz, Linz
  - Salzburg Regional Hospital, Salzburg
  - Hanusch Hospital, Vienna
  - Medical University Vienna, Vienna
  - Hospital Wels-Grieskirchen, Wels
- Belgium (4):
  - Centre du Cancer et D'hematologie, Brussels
  - UZA, Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
  - Haematolgy, University of Liège, Liège
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv
  - Specialized Hospital for Active Treatment of Hematological Diseases, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
  - Multiprofile Hospital for Active Treatment - Hristo Botev, Vratsa, First Department of Internal Medicine, Vratsa
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Institute of Hematology and Blood Transfusion, Prague
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
- France (3):
  - Institute Paoli-Calmettes, Marseille
  - Hospital Saint-Louis, Paris
  - Clinical Research Center CIC, Poitiers
- Germany (3):
  - Aachen University Hospital, Medical Clinic IV, Aachen
  - University Hospital Bonn, Center for Internal Medicine, Medical Clinic and Outpatient Clinic III, Bonn
  - University Hospital Carl Gustav Carus, Medical Clinic and Polyclinic I, Dresden
- Hungary (5):
  - St Istvan and St Laszlo Hospital of Budapest, Budapest
  - University of Debrecen, Debrecen
  - Bekes County Pandy Kalman Hospital, 1st Department of Medicine, Hematology, Gyula
  - Kaposi Mor County Teaching Hospital, Kaposvár
  - University of Szeged, Albert Szent-Gyorgyi Clinical Center, Koranyi fasor 6, Szeged
- Italy (2):
  - Careggi University Hospital, Florence
  - Foundation IRCCS Policlinico San Matteo, Pavia
- Poland (6):
  - Andrzej Mielecki Independent Public Clinical Hospital of Medical University of Silesia in Katowice, Katowice
  - University Hospital in Cracow, Krakow
  - Independent Public Teaching Hospital No.1 in Lublin, Lublin
  - Fryderyk Chopin Provincial Specialized Hospital, Rzeszów
  - Nicolaus Copernicus Municipal Specialist Hospital, Torun
  - Institute of Hematology and Transfusion Medicine, Warsaw
- Romania (4):
  - Emergency Clinical County Hospital Brasov, Brasov
  - Bucharest University Emergency Hospital, Bucharest
  - Coltea Clinical Hospital, Bucharest
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Cluj-Napoca
- Russia (6):
  - Baranov Republican Hospital, Petrozavodsk
  - First Pavlov State Medical University of St. Petersburg, Saint Petersburg
  - Samara Kalinin Regional Clinical Hospital, Samara
  - Komi Republican Oncology Center, Syktyvkar
  - Tula Regional Clinical Hospital, Tula
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- Slovakia (2):
  - University Hospital with Outpatient Clinic F.D. Roosevelt, Banská Bystrica
  - Saint Cyril and Metod University Hospital Bratislava, Bratislava
- Spain (2):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
- Ukraine (5):
  - Cherkasy Regional Oncology Center, Regional Treatment and Diagnostics Hematology Center, Cherkasy
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Dnipropetrovsk
  - National Research Center for Radiation Medicine, Institute of Clinical Radiology, Kiev
  - Institute of Blood Pathology and Transfusion Medicine, Lviv
  - O.F. Herbachevskyi Regional Clinical Hospital, Zhytomyr

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verger E, Soret-Dulphy J, Maslah N, Roy L, Rey J, Ghrieb Z, Kralovics R, Gisslinger H, Grohmann-Izay B, Klade C, Chomienne C, Giraudier S, Cassinat B, Kiladjian JJ. Ropeginterferon alpha-2b targets JAK2V617F-positive polycythemia vera cells in vitro and in vivo. Blood Cancer J. 2018 Oct 4;8(10):94. doi: 10.1038/s41408-018-0133-0. PMID 30287855